CLINICAL TRIAL: NCT06589089
Title: Prospective Study of Autologous Hematopoietic Stem Cell Boost to Improve Myelosuppression in B-NHL Patients with High-risk Immunologic Hematologic Toxic After Chimeric Antigen Receptor T-Cell Immunotherapy
Brief Title: Autologous Hematopoietic Stem Cell Boost Study After CAR-T Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Prof., Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-SCB
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients treated with stem cell boost (Experimental): If the patient continues to have unrelieved hematologic toxicity after CAR-T cell therapy, consider infusing a reserve of stem cells; If there is no significant recovery from myelosuppression, another stem cell infusion can be performed.
  Interventions: Drug: autologous hematopoietic stem cell

INTERVENTIONS:
Drug: autologous hematopoietic stem cell — Intervention were given myelosuppression occurring that cannot be controlled with other drugs as judged by the investigators

SUMMARY:
This is a prospective, single-arm, open study to observe the efficacy and safety of the CART-SCB regimen (Clinical Regimen for the Prospective Study of Autologous Hematopoietic Stem Cell Boost for the Improvement of Bone Marrow Suppression in Patients with High-Risk Immunohematologic Toxicity Lymphoma After Chimeric Antigen Receptor T (CAR-T)-Cell Immunotherapy Therapy) . After the patient has completed CAR-T therapy, if the patient has unrelieved hematologic toxicity, consider infusing a reserve of stem cells; if myelosuppression has not been significantly relieved, stem cell infusion can be performed again.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and gender-neutral;
* Diagnosis of B-cell non-Hodgkin lymphoma confirmed histologically or cytologically according to World Health Organization 2016 criteria;
* Prior CAR-T cell immunotherapy;
* Patients who are at high risk according to the CAR-HEMATOTOX score prior to leukapheresis; or patients who are clinically considered potentially at high risk for hematologic toxicity following immunotherapy (including age ≥60 years; or Eastern Cooperative Oncology Group (ECOG) Performance Status≥ 2 points; or number of prior lines of therapy ≥ 2, etc.);
* Myelosuppression as determined by the investigator has occurred after CAR-T therapy;
* Have a storage of stem cell;
* Stable lymphoma disease status (final investigator-assessed efficacy CR/PR);
* Bone marrow biopsy to rule out hemophilia/infection/bone marrow infiltration;
* Adequate organ function;
* Able to provide written informed consent (ICF) and able to understand and agree to comply with the study requirements and assessment schedule;
* Patients of childbearing potential must be willing to use highly effective contraception for the duration of the study, and for 120 days after the last dose of treatment.

Exclusion Criteria:

* History of allogeneic hematopoietic stem cell transplantation;
* History of epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the central nervous system;
* Presence of or current concurrent other malignancies within the past 2 years, with the exception of cured carcinoma in situ of the uterine cervix, non-melanoma skin cancers, and superficial bladder tumors (Ta (non-invasive tumors), Tis (carcinoma in situ), and T1 (tumors infiltrating the basement membrane));
* Suffering from severe cardiovascular disease: grade II or greater myocardial ischemia or myocardial infarction, poorly controlled arrhythmias; grade III-IV cardiac insufficiency according to New York Heart Association (NYHA) criteria, or cardiac ultrasound suggestive of a left ventricular ejection fraction (LVEF) <50%;
* Allergy to any investigational drug or excipient;
* Presence of any active autoimmune disease (including, but not limited to: autoimmune hepatitis, interstitial pneumonitis, uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism), or known history of allograft transplantation, or patients with prolonged and heavy use of hormones or use of other immune-modulating agents or other patients who, as assessed by the Investigator Patients who are considered to have an impact on study treatment;
* Have an active infection;
* History of uncontrolled systemic disease, including diabetes mellitus, hypertension, and acute pulmonary disease;
* Known human immunodeficiency virus (HIV) infection;
* Presence of an underlying medical condition or alcohol/substance abuse or dependence that is not conducive to the administration of study medication, or that may interfere with the interpretation of results, or that puts the patient at high risk for developing treatment complications;
* End-organ damage due to autoimmune disease (e.g., Crohns disease, rheumatoid arthritis, systemic lupus erythematosus) within the past 2 years, or the need for systemic immunosuppression or other systemic disease-control medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
1-year overall survival | 1 year after CAR-T cell infusion
  Overall survival was defined as the time from the date of leukapheresis to the date of death from any cause.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | End of treatment visit (1 years after stem cell infusion)
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Best objective response rate | End of treatment visit (1 years after stem cell infusion)
  Defined as the proportion of patients with an efficacy evaluation of complete response (CR) or partial response (PR) at any time point after infusing back CAR-T cells as a percentage of all patients, with efficacy assessed by the investigators according to the 2014 Lugano efficacy criteria
Best complete response rate | End of treatment visit (1 years after stem cell infusion)
  Defined as the proportion of patients with an efficacy evaluation of CR at any time point after infusing back CAR-T cells as a percentage of all patients, with efficacy assessed by the investigators according to the 2014 Lugano efficacy criteria
Time to reponse | End of treatment visit (1 years after stem cell infusion)
  Time from CAR-T cell infusion to the first assessment of CR or PR on the basis of investigator assessments according to 2014 Lugano criteria.
Duration of response | End of treatment visit (1 years after stem cell infusion)
  Time from the first efficacy assessment of CR or PR to the time of first disease progression on the basis of investigator assessments according to 2014 Lugano criteria.
Progression-free survival | End of treatment visit (1 years after stem cell infusion)
  Progression-free survival was defined as the time from the date of leukapheresis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | End of treatment visit (1 years after stem cell infusion)
  Overall survival was defined as the time from the date of leukapheresis to the date of death from any cause.
Overall days of hospitalization | End of treatment visit (1 years after stem cell infusion)
  Defined as total number of days admitted to the hospital since being infused back for CAR-T, including days of readmission for supportive care for myelosuppression

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China